CLINICAL TRIAL: NCT00754182
Title: Comparison of Esthetic Results Between Subcuticular Suture and Synthetic Glue in Thyroidectomy Incision: a RCT
Brief Title: Subcuticular Suture Versus Synthetic Glue in Thyroidectomy Incision
Acronym: SCSvsSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Matteo Alicandri-Ciufelli, U.O.C. Otorinolaringoiatria Azienda Ospedaliero-Univeritaria di Modena
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2454/C.E.
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2009-03

CONDITIONS: Goiter; Thyroid Neoplasms; Parathyroid Pathologies
Keywords: thyroidectomy; surgery; synthetic glue; subcuticular suture
MeSH Terms: conditions — Goiter; Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients underwent thyroidectomy, emithyroidectomy, parathyroidectomy sutured with synthetic glue
  Interventions: Device: Octylcyanoacrylate (Dermabond)
- B (Active Comparator): Patients underwent thyroidectomy, emithyroidectomy, parathyroidectomy sutured with subcuticular suture
  Interventions: Device: Subcuticular reabsorbable suture (Caprosyn)

INTERVENTIONS:
Device: Octylcyanoacrylate (Dermabond) — Synthetic glue for surgical use (skin closure)
  Other Names: Dermabond
  Arms: A
Device: Subcuticular reabsorbable suture (Caprosyn) — Every stitch is positioned in the subcuticular tissue by a continuous technique
  Other Names: Caprosyn
  Arms: B

SUMMARY:
The aim of this study is to compare aesthetic results of two different type of sutures (subcuticular versus synthetic glue) in post-thyroidectomy incisions. It is a randomized clinical trial (single blinded) designed as a superiority study, since in the authors' hypotheses glue can give better results compared with subcuticular suture in this particular district. Secondary objective is to investigate if other factors (like the use of cold/warm blade, the sex, the presence of diabetes, the lenght of incision) can influence aesthetic results.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent thyroidectomy, emithyroidectomy, parathyroidectomy

Exclusion Criteria:

* Former neck operations with external incisions
* Post-operative bleeding
* Cervical nodes involvement (with the necessity of widened incisions)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Scar evaluation scale for short term esthetic results (Hollander, J. E., Singer, A. J., Valentine, S., and Henry, M. C. Wound registry: Development and validation. Ann. Emerg. Med. 25: 675, 1995.) | 10 days

SECONDARY OUTCOMES:
Scar Evaluation Scale (by Adam J. Singer, M.D. et al. "Development and Validation of a Novel Scar Evaluation Scale" Plastic and Reconstructive Surgery ,December 2007 Volume 120, Number 7 ,1892-1897) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Alicandri-Ciufelli, MD, Principal Investigator — Otorinolaringoiatria, Policlinico di Modena
Locations (1):
- Policlinico di Modena, Modena, Modena, Italy